CLINICAL TRIAL: NCT00796952
Title: Muscle Composition and Function for Swallowing in Head/Neck Cancer Patients Undergoing Radiotherapy: a Randomized Controlled Trial of Swallowing Therapy"
Brief Title: Muscle Composition and Function for Swallowing in Head/Neck Cancer Patients
Acronym: Pharyngocise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM009
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Head & Neck Cancer
Keywords: Head/ neck cancer; Swallowing; behavioral treatment
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (Active Comparator): Patient management by the attending Radiation oncologist "as usual".
  Interventions: Behavioral: focused attention sessions
- Pharyngocise (Experimental): Standardized high intensity behavioral swallowing therapy (Pharyngocise) comprised a battery of direct isometric / isotonic exercises and appropriate dietary modification, under the direction of the study speech pathologist, twice daily for the duration of the patient's total course of their chemo-radiation treatment (up to a maximum of 6 weeks)
  Interventions: Behavioral: Pharyngocise
- Valchuff (Sham Comparator): Standardised sham swallowing therapy comprised a buccal extension maneuver ("valchuff") and appropriate dietary modification, under the direction of the study speech pathologist, twice daily each week for the duration of the patient's total course of chemo-radiation treatment.
  Interventions: Behavioral: Valchuff

INTERVENTIONS:
Behavioral: focused attention sessions — Patient management by the attending Radiation oncologist "as usual". Patients assigned to this condition received focused attention sessions during the total course of their CRT treatment from a Speech Language Pathologist, consisting of weekly phone calls to monitor their swallowing outcome during the radiotherapy period.
  Arms: Usual Care
Behavioral: Valchuff — Standardised sham or placebo swallowing therapy comprised a buccal extension maneuver ("valchuff") and appropriate dietary modification, under the direction of the study speech pathologist, twice daily each week for the duration of the patient's total course of CRT treatment.
  Arms: Valchuff
Behavioral: Pharyngocise — Standardized high intensity behavioral swallowing therapy (Pharyngocise) comprised a battery of direct isometric / isotonic exercises and appropriate dietary modification, under the direction of the study speech pathologist, twice daily for the duration of the patient's total course of their CRT treatment (up to a maximum of 6 weeks)
  Arms: Pharyngocise

SUMMARY:
Swallowing dysfunction after chemo-radiation is common, but there is no reliable evidence for how it should be managed. This pilot randomized controlled trial evaluated the relative benefit of a battery of isometric / isotonic exercises on the maintenance of muscle composition and function for swallowing in Head / Neck Cancer patients undergoing chemo-radiation therapy.

DETAILED DESCRIPTION:
Swallowing deficits resulting from oropharyngeal cancer and the ablative therapies used to control the disease are often devastating to the functional feeding outcome in these patients. Most patients will experience some degree of dysphagia along with nutritional decline. In particular, the swallowing outcome of those patients treated with external beam radiation is suggested to be poorer than those patients treated by surgical interventions alone. It has also been postulated that the formation of radiation-induced fibrotic tissue, along with the acute radiation effects (edema, mucositis, xerostomia) may act collectively to promote muscular disuse or atrophy, and the noted decline in swallowing function. We therefore suggest that a program of swallowing exercises may help facilitate and maintain muscle function in the oral cavity and pharynx during radiotherapy, thus preserving or supporting swallowing function in these patients.

This study will follow a randomized controlled trial design. Patients with confirmed head / neck cancer identified for planned radiotherapy will undergo a baseline evaluation including clinical and instrumental swallowing assessment, nutritional examination, and MRI prior to CRT. Subjects will then be randomized to one of three intervention arms representing control, placebo and intervention groups. Patients will be treated for 6 weeks and progress reassessed at 6 months. Outcome assessment will be completed by a blinded observer. Primary outcomes include; I)Oropharyngeal active muscle volume, signal intensity, and tissue composition over time as identified by T2 weighted MRI, II)Level of functional swallowing ability,III)Patient perception of swallowing function and quality of life.The results of the study will provide information on the efficacy (or lack of efficacy) of isometric / isotonic exercises for the maintenance of swallowing function post radiotherapy for Head /Neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Head / neck cancer of the oropharyngeal or adjacent regions, confirmed by clinical history and exam, with positive cross sectional imaging studies and histopathological biopsy excluding other pathology.
* Planned to undergo external beam radiation therapy,
* No previous history of nonoral feeding for cancer related illness,
* Able to undergo MRI procedures.
* Physician / patient agreement to participate

Exclusion Criteria:

* Planned surgical intervention
* Existence of a co-existing neurological or medical disorder known to cause dysphagia
* Prior radiotherapy or surgery to the head / neck region that could contribute to dysphagia.
* Previous swallowing therapy within four weeks of randomization

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2001-11; Primary Completion 2004-07 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal muscle volume and signal intensity measured by T2 weighted MRI | Baseline, 6 weeks( end of CRT), 6 months(following CRT)
Level of functional swallowing ability- measured by functional eating score (FOIS), clinical swallowing score, videoendoscopy and videofluoroscopic evaluation | Baseline, 6 week(end of CRT), 6 months(following CRT)
Patient perception of swallowing ability | Baseline, 6 weeks (end of CRT), 6 months (following CRT)
Quality of Life | Baseline, 6 weeks (end of CRT), 6 months (following CRT)

SECONDARY OUTCOMES:
Taste perception | Baseline, 6 weeks (end of CRT), 6 months (following CRT)
Perception of smell | Baseline, 6 weeks (end of CRT), 6 months (following CRT)
Salivation rates | Baseline, 6 weeks (end of CRT), 6 months (following CRT)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Carnaby-Mann, PhD, Principal Investigator — University of Florida; Michael Crary, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Health Science Center, Gainesville, Florida, United States